CLINICAL TRIAL: NCT02843516
Title: Detection Rate of Atrial Fibrillation in Patients Implanted With ILRs
Status: Completed | Type: Observational
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Peter J Pugh, Consultant Cardiologist, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: 190674
Record Dates: First submitted 2016-06-28; First posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients with stroke: patients with stroke
  Interventions: Other: No intervention
- patients without stroke: patients without stroke
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Implantable Loop Recorders (ILRs), are subcutaneous heart monitors, which are implanted for different reasons including syncope (fainting), pre syncope (near fainting), palpitations and stroke. They monitor the heart and detect abnormalities.

Atrial fibrillation (irregular heart rhythm),is a common cardiac arrhythmia associated with a five-fold risk of stroke. Atrial Fibrillation increases the risk of stroke in patients to a different degree according to a risk stratification score. Anticoagulation is recommended to all high-risk patients.

Recent published studies have shown a high incidence of Atrial Fibrillation detected by ILRs in patients with previous stroke.

It is not known whether a similar incidence of Atrial Fibrillation occurs in patients without previous stroke. It is also not know ''how much'' Atrial Fibrillation is necessary to increase the risk of stroke, how relevant the finding of Atrial Fibrillation is and whether everybody with Atrial Fibrillation should have anticoagulation or whether a "bit of Atrial Fibrillation" is actually normal in most people.

The purpose of this study is to identify and compare the rate and the burden of Atrial Fibrillation (more or less than 30 seconds) in patients with and without previous stroke.

Medical notes and Implantable Loop Recorder records of the patients that had the devices implanted in Addendbrooke's Hospital from March 2009 up to 1 month after the implantation of the latest device will be inspected in order to identify whether the device had detected Atrial Fibrillation and if so the burden of Atrial Fibrillation in the two different groups of patients (with and without previous stroke).

The risk of stroke for each patient will be calculated. Echocardiographic (ultrasound scan of the heart)risk factors for Atrial Fibrillation will be identified and compared between the two groups.

This is going to be a retrospective study and we will be inspecting patients' data only.

DETAILED DESCRIPTION:
Implantable Loop Recorders (ILRs), are subcutaneous heart monitors, which are implanted for different reasons including syncope (fainting), pre syncope (near fainting), palpitations and stroke. They monitor the heart and detect abnormalities.

Atrial fibrillation (irregular heart rhythm),is a common cardiac arrhythmia associated with a five-fold risk of stroke. Atrial Fibrillation increases the risk of stroke in patients to a different degree according to a risk stratification score. Anticoagulation is recommended to all high-risk patients.

Recent published studies have shown a high incidence of Atrial Fibrillation detected by ILRs in patients with previous stroke.

It is not known whether a similar incidence of Atrial Fibrillation occurs in patients without previous stroke. It is also not know ''how much'' Atrial Fibrillation is necessary to increase the risk of stroke, how relevant the finding of Atrial Fibrillation is and whether everybody with Atrial Fibrillation should have anticoagulation or whether a "bit of Atrial Fibrillation" is actually normal in most people.

The purpose of this study is to identify and compare the rate and the burden of Atrial Fibrillation (more or less than 30 seconds) in patients with and without previous stroke.

Medical notes and Implantable Loop Recorder records of the patients that had the devices implanted in Addendbrooke's Hospital from March 2009 up to 1 month after the implantation of the latest device will be inspected in order to identify whether the device had detected Atrial Fibrillation and if so the burden of Atrial Fibrillation in the two different groups of patients (with and without previous stroke).

The risk of stroke for each patient will be calculated. Echocardiographic (ultrasound scan of the heart)risk factors for Atrial Fibrillation will be identified and compared between the two groups.

This is going to be a retrospective study and we will be inspecting patients' data only..

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged 18 years or above.
* Patients with Implantable Loop Recorder

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients implanted with Implantable Loop Recorders from March 2009 up to 1 month (first follow up) of the latest ILR implantation.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2009-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Atrial Fibrillation in patients with and without previous stroke | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pugh, MBBS, MRCP, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No